CLINICAL TRIAL: NCT06112171
Title: Performance of the Shockwave Medical Peripheral Lithotripsy System vs Standard Balloon Angioplasty for Lesion Preparation Prior to Supera Stent Implantation in the Treatment of Symptomatic Severely Calcified Femoropopliteal Lesions in PAD
Brief Title: Comparison of a Lithotripsy vs Standard Preparation Followed by Stenting With Supera Stent in Femoropopliteal Lesions
Acronym: CRACK-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP_23/001
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Calcification; Lithotripsy
MeSH Terms: conditions — Peripheral Arterial Disease; Calcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular lithotripsy arm (Other): Treatment with Lithotripsy system followed by Supera stent implantation in lesion segments with severe calcification.
  Interventions: Procedure: Intravascular lithotripsy
- Standard lesion preparation arm (Other): Treatment with Balloon angioplasty with a conventional and/or high-pressure balloon angioplasty followed by Supera stent implantation in lesion segments with severe calcification.
  Interventions: Procedure: Standard lesion preparation

INTERVENTIONS:
Procedure: Intravascular lithotripsy — Lesion preparation with Shockwave Medical Peripheral Lithotripsy System
  Arms: Intravascular lithotripsy arm
Procedure: Standard lesion preparation — Lesion preparation with Standard and/or High-Pressure Balloon Angioplasty
  Arms: Standard lesion preparation arm

SUMMARY:
This study is an investigator-initiated, prospective, single-center, 1:1 randomized pilot study.

The trial evaluates the safety and efficacy of intravascular lithotripsy in comparison to standard lesion preparation using standard and/or high-pressure balloon angioplasty in patients with femoropopliteal artery disease. All patients will receive subsequent Supera stent implantation at the operator's discretion. Additional standard nitinol bare metal stent (BMS), drug-eluting stent or covered stent implantation is at the operator's discretion.

Patients will be stratified for total occlusions.

DETAILED DESCRIPTION:
All enrolled subjects will be followed up through 60 months. At 6, 12, 24, 36 MFU after index procedure the incidence of restenosis will be assessed by DUS.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥ 18
* Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved inform consent form
* Subject understands the duration of the study, agrees to attend follow-up visits, and agrees to complete the required testing
* Rutherford Classification 2-5
* Subject has a de novo or restenotic lesion in SFA and/or PPA not exceeding the medial femoral epicondyle with ≥ 70% stenosis documented angiographically
* No previous stent in the target lesion, if target vessel was previously stented the stent should be at least 3cm apart
* Target lesion length is ≥ 10cm, no maximum lesion length limit
* Severe calcification on fluoroscopy defined by PACSS Grade 4: 1) bilateral calcification and 2) extending ≥50mm in length
* Multiple lesions with max. 3cm healthy vessel segment in between lesions can be considered at the discretion of the operator as one lesion
* Reference vessel diameter (RVD) ≥ 4 mm and ≤ 6.5 mm by visual estimation
* Patency of at least one infrapopliteal artery to the ankle (< 50% diameter stenosis) in continuity with the native femoropopliteal artery
* A guidewire has successfully traversed the target treatment segment (both intraluminal and subintimal crossing allowed)

Exclusion Criteria:

* Failure to successfully cross the target lesion
* Presence of fresh thrombus in the lesion
* Presence of aneurysm in the target vessel/s
* Presence of a stent in the target lesion, at least 3cm from any previously stent in target vessel
* Prior vascular surgery of the target lesion
* Stroke or heart attack within 3 months prior to enrollment
* Enrolled in another investigational drug, device or biologic study that has not reached the primary endpoint
* Life expectancy of less than one year
* Known allergies or sensitivity to heparin, aspirin, other anticoagulant/ antiplatelet therapies or contrast media that cannot be adequately pre-treated prior to index procedure
* Rutherford Classification of 0, 1, or 6
* Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
* Receiving immunosuppressant therapy
* Pregnant or breast-feeding females
* History of major amputation (defined as amputation above ankle joint) in the same limb as the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy | During the Procedure
  Procedural success defined as residual stenosis ≤ 30% without flow-limiting dissection (≥Grade D) in the final angiogram and without the need of additional stent implantation.
Rate of primary outcome events | 12 month
  Composite endpoint defined as freedom from device and procedure-related death, freedom from both target limb major amputation and clinically-driven target lesion revascularization

SECONDARY OUTCOMES:
Rate of vessel rupture | During the Procedure
  Rate of vessel rupture
Need of additional stent implantation | During the Procedure
  Need of additional stent implantation
Procedure Time (min) | During the Procedure
  Procedure Time (min)
Fluoroscopy Duration (min) | During the Procedure
  Fluoroscopy Duration (min)
Radiation dose area product | During the Procedure
  Radiation dose area product
Additional need of intra-procedural pain medication | During the Procedure
  Additional need of intra-procedural pain medication
Perception of procedural pain evaluated using a numerical rating scale from 0 (no pain) to 10 (severest pain) | During the Procedure
  Perception of procedural pain evaluated using a numerical rating scale from 0 (no pain) to 10 (severest pain)
Rate of any dissections after lesion preparation and in the final angiogram | During the Procedure
  Rate of any dissections after lesion preparation and in the final angiogram
Rate of primary patency | 6, 12, 24 and 36 months
  Rate of primary patency
Rate of Duplex-defined binary restenosis (PVR >2.4) of the target lesion | post-procedure until discharge from hospital (up to 48 hours) and at 6, 12, 24 and 36 months or at any time of re-intervention
  Rate of Duplex-defined binary restenosis (PVR >2.4) of the target lesion
Rate of Clinically-driven Target lesion revascularization | 30 days, 6, 12, 24, 36, 48 and 60 months
  Rate of Clinically-driven Target lesion revascularization
Rate of Freedom from Major Adverse Event (defined as death, Target lesion revascularization, Target vessel revascularization and target limb major amputation) | 30 days, 6, 12, 24, 36, 48 and 60 months
  Rate of Freedom from Major Adverse Event (defined as death, Target lesion revascularization, Target vessel revascularization and target limb major amputation)
Rate of All-cause mortality | 30 days, 6, 12, 24, 36, 48 and 60 months
  Rate of All-cause mortality
Ankle-brachial index (ABI) | 6, 12, 24 and 36 months
  The ABI is calculated by dividing the highest of the dorsalis pedis and posterior tibial pressures in each leg by the highest of the brachial pressures.
  Value less than 0.90 indicates a diagnosis of PAD.
Rutherford Classification | 6, 12, 24 and 36 months
  Rutherford Classification Scale from 0=Asymptomatic, 1=Mild claudication, 2=Moderate claudication, 3=Severe claudication, 4=Ischemic rest pain, 5=Minor tissue loss up to worst classification 6=Major tissue loss
Walking Impairment Questionnaire (WIQ) | 6, 12, 24 and 36 months
  The products are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (representing the inability to perform any of the tasks) to 100 (representing no difficult with any of the tasks).
EQ-5D-5L questionnaire | 6, 12, 24 and 36 months
  The EQ-5D-5L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: o problems, slight problems, moderate problems, severe problems and extreme problems.
EQ VAS | 6, 12, 24 and 36 months
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 100% 'Best imaginable health state' and 0% 'Worst imaginable health state'.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Steiner, Prof. Dr., Principal Investigator — University Leipzig
Locations (1):
- University Clinic Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No